CLINICAL TRIAL: NCT03271593
Title: Impact of Rotavirus Vaccination on Hospital Pressures at a Large Paediatric Hospital in the UK: an Ecological Study
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 205369
Record Dates: First submitted 2016-08-05; First posted 2017-09-05 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Gastroenteritis
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All children admitted: All children admitted to hospital
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The impact of rotavirus vaccination on the burden of disease has been well documented. However, the anticipated reduction in hospital pressures has yet to be described. This study will provide quantitative measures of hospital pressure prior to and post vaccine introduction, provide a template for future hospital pressures studies related to vaccine introduction and provide measures which could be used in an economic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* All children aged ≤15 years being hospitalised (with overnight stay or day clinic) for whatever reason during the study period

Exclusion Criteria:

* None

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children <15 years admitted to Alder Hey Children's NHS Foundation Trust. Four sub-populations: All admissions for any cause; Admission for an infectious disease; Admission for all cause gastroenteritis; Admission for Rotavirus gastroenteritis
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-09-23 (Actual)

PRIMARY OUTCOMES:
Change in bed day occupancy (BDO) rates | During the study observation period of 15 years (1st July 2000 - 30th June 2015)
  BDO rate is measured as the number of bed days occupied divided by the total number of bed days available in a ward during a fixed time period. BDO rate will be measured in overall admissions, admissions for infectious disease only, admissions for gastro-enteritis only, admissions for rotavirus induced gastro-enteritis only
Change in turnover (TO) rates | During the study observation period of 15 years (1st July 2000 - 30th June 2015)
  TO rate is the change in average hospital duration measured as average number of days stay per admission. TO rate will be measured in overall admissions, admissions for infectious disease only, admissions for gastro-enteritis only, admissions for rotavirus induced gastro-enteritis only
Change in early unplanned readmission (UR) rates | During the study observation period of 15 years (1st July 2000 - 30th June 2015)
  UR rate (within 7 days after discharge) is measured as the number of readmissions ≤7 days after discharge (x100) divided by the total number of discharges. UR rate will be measured in overall admissions, admissions for infectious disease only, admissions for gastro-enteritis only, admissions for rotavirus induced gastro-enteritis only
Change in rate of nosocomial infections (NOSO) | During the study observation period of 15 years (1st July 2000 - 30th June 2015)
  NOSO rate is measured as positive test from a test taken >2 days after admission. NOSO rate will be measured in overall admissions, admissions for infectious disease only, admissions for gastro-enteritis only, admissions for rotavirus induced gastro-enteritis only
Change in number of rotavirus gastroenteritis (RVAG) tests taken | During the study observation period of 15 years (1st July 2000 - 30th June 2015)
  RVAG rate will be measured in overall admissions, admissions for infectious disease only, admissions for gastro-enteritis only, admissions for rotavirus induced gastro-enteritis only
Change in number of positive test results | During the study observation period of 15 years (1st July 2000 - 30th June 2015)
  Number of positive RVAG test results will be measured in overall admissions, admissions for infectious disease only, admissions for gastro-enteritis only, admissions for rotavirus induced gastro-enteritis only
Change in rate of hospitalization in children less that 5 years old | During the study observation period of 15 years (1st July 2000 - 30th June 2015)
  Change in rate of hospitalization (in children less that 5 years old) will be measured in overall admissions, admissions for infectious disease only, admissions for gastro-enteritis only, admissions for rotavirus induced gastro-enteritis only

SECONDARY OUTCOMES:
Development of a Quality of Care (QoC) score | During the study observation period of 15 years (1st July 2000 - 30th June 2015)
  To develop the QoC score, a baseline rate/score for each outcome measure out-of-season (June-December) will be developed pre-vaccine introduction (vaccine introduction: 30th July 2013). Each outcome measure in the pre-vaccine period and post-vaccine period in-peak-season (January to May) will be scaled against that score. An overall QoC-Score pre- and post-vaccine in peak season will be calculated by summing scores for each outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Heinsbroek E, Hungerford D, Cooke RPD, Chowdhury M, Cargill JS, Bar-Zeev N, French N, Theodorou E, Standaert B, Cunliffe NA. Do hospital pressures change following rotavirus vaccine introduction? A retrospective database analysis in a large paediatric hospital in the UK. BMJ Open. 2019 May 15;9(5):e027739. doi: 10.1136/bmjopen-2018-027739. PMID 31097487
- Available data/document: Clinical Study Report — https://www.gsk-clinicalstudyregister.com/study/205369?search=study&search_terms=205369#csr — Results disclosed in the Clinical Study Report.